CLINICAL TRIAL: NCT01900587
Title: A Single-Dose, Open-Label, Randomized, 2-Way Crossover Pivotal Study to Assess Bio-equivalence of a New Tapentadol Extended-Release (TRF) 50-mg Tablet With Respect to a Tapentadol Extended-Release (PR2) 50-mg Tablet Under Fasted Conditions in Healthy Subjects
Brief Title: A Pivotal Study to Evaluate the Bio-equivalence of the Tapentadol Extended-Release (ER) Tamper-resistant Formulation (TRF) Tablet to the Current Tapentadol ER Prolonged-release 2 (PR2) Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR100456; R331333-PAI-1059
Record Dates: First submitted 2013-07-12; First posted 2013-07-16 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
Keywords: Healthy; Bio-equivalence; Tapentadol extended release; Tamper-resistant formulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tapentadol Extended release (ER) TRF then tapentadol ER PR2 (Experimental): Single dose of tapentadol ER 50 milligram (mg), tamper-resistant formulation (TRF) tablet will be administered under fasted condition in first treatment period; after that in second treatment period, single-dose of tapentadol ER 50 mg, prolonged released (PR2) tablet will be administered under fasted condition. A washout period of 7 to 14 days will be maintained between each treatment period.
  Interventions: Drug: Tapentadol ER Tamper-resistant Formulation (TRF); Drug: Tapentadol ER Prolonged-Release 2 (PR2)
- Tapentadol ER PR2 then tapentadol ER TRF (Experimental): Single dose of tapentadol ER 50 milligram (mg), PR2 tablet will be administered under fasted condition in first treatment period; after that in second treatment period, single-dose of tapentadol ER 50 mg, TRF tablet will be administered under fasted condition. A washout period of 7 to 14 days will be maintained between each treatment period.
  Interventions: Drug: Tapentadol ER Tamper-resistant Formulation (TRF); Drug: Tapentadol ER Prolonged-Release 2 (PR2)

INTERVENTIONS:
Drug: Tapentadol ER Tamper-resistant Formulation (TRF) — Single dose of tapentadol ER 50 milligram (mg), will be administered under fasted condition.
Drug: Tapentadol ER Prolonged-Release 2 (PR2) — Single dose of tapentadol ER 50 milligram (mg), prolonged release tablet will be administered under fasted condition.

SUMMARY:
The purpose of this study is to evaluate bio-equivalence of tapentadol extended-release (ER) tamper-resistant formulation (TRF) tablet, to the current tapentadol ER, prolonged-release formulation 2 (PR2) tablet, in healthy participants.

DETAILED DESCRIPTION:
This is a single-dose, open-label (a medical research study in which participants and researchers are told which treatments the participants are receiving, "unblinded"), single-centre, randomized (like the flip of a coin; 50/50 chance of receiving a study treatment), and 2-way crossover (groups of participants receive two or more interventions in a particular order) study of a single-dose tapentadol in healthy participants under fasted conditions. The study consists of 3 parts: Screening (2 to 21 days before the study commences), Open-label Treatment (single-dose treatment on Day 1 of each period separated with wash-out period of 7 to 14 days) and End of study (Day 3 of treatment Period 2). The duration of participation in the study for an individual participant will be up to 5.5 weeks (including Screening). Participants will be randomly assigned to one of the 2 treatment sequence groups. Participants assigned to the first treatment sequence will receive tapentadol TRF 50 milligram (mg) tablet, and after a washout period, participants will receive tapentadol PR2 50-mg tablet. Participants assigned to the second treatment sequence will receive tapentadol PR2 50-mg tablet, and after washout period, participants will receive tapentadol TRF 50-mg tablet. Bio-equivalence will be primarily evaluated by pharmacokinetics parameters. Participant's safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants deemed healthy on the basis of pre-study physical examination, medical history (including smoking habits), 12-lead electrocardiogram (ECG), vital signs, and clinical laboratory parameters (serum chemistry, serology and hematology) performed within 21 days before study drug administration
* Female participants must be post-menopausal, surgically sterile, or, if of childbearing potential/sexually active, be practicing an effective method of birth control throughout the study. Women must have a negative serum beta human chorionic gonadotropin pregnancy test at Screening and on Day -1 of each treatment period. Men must not impregnate their partners
* Participants with body mass index (BMI) (weight [kilogram {kg}]/height [meter {m}^2]) in-between 20 to 28 kg/m^2, inclusive, and body weight not less than 50 kg
* Participants with blood pressure between 100 and 140 millimeters of mercury (mmHg) systolic, inclusive, and between 50 and 90 mmHg diastolic
* Participants who smokes no more than 10 cigarettes, or 2 cigars, or 2 pipes of tobacco per day for at least 6 months before the first study drug administration

Exclusion Criteria:

* Participants with history of seizure disorder or epilepsy or mild or moderate traumatic brain injury, stroke, transient ischemic attack, or brain neoplasm within 1 year of screening, or severe traumatic brain injury within 15 years of screening, or severe traumatic brain injury resulting in ongoing squealed suggesting transient changes in consciousness or symptoms
* Participants with history of a gastrointestinal disease affecting absorption, gastric surgery or history of or current significant medical illness including cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders, lipid abnormalities, significant pulmonary disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the Investigator considers should exclude the participants
* Participants who received an experimental drug or used an experimental medical device within 30 days or within a period less than 10 times the drug's half-life, whichever is longer, before the first dose of the study drug is scheduled or to participate in an investigational drug study for at least 60 days after completion of the study
* Participants who have positive test for drugs of abuse, such as cannabinoids, alcohol, opiates, cocaine, amphetamines, benzodiazepines, or barbiturates at Screening or Day -1 of each treatment period
* Participants who donated blood or blood products or had substantial loss of blood (greater than 500 milliliter) within 2 months before the first administration of study drug

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2010-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Maximum Serum Concentration (C[max]) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36 and 48 hours post-dose of study medication
  The C(max) is the maximum serum concentration which will be observed at the defined time points.
Area Under the Serum Concentration-Time Curve From Time Zero to Infinite Time (AUC [infinity]) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36 and 48 hours post-dose of study medication
  The AUC (infinity) is the area under the serum concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z), wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time; and C(last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.
Area Under the Serum Concentration-Time Curve From Time Zero to Infinite Time (AUC [last]) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36 and 48 hours post-dose of study medication
  The AUC (last) is the area under the serum concentration-time curve from time zero time of the last quantifiable concentration C(last), and C(last) is the last observed quantifiable concentration.

SECONDARY OUTCOMES:
Time to Reach the Maximum Serum Concentration (T[max]) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36 and 48 hours post-dose of study medication
  The T[max] is time to reach the observed maximum serum concentration.
Percentage of AUC(infinity) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36 and 48 hours post-dose of study medication
  Percentage of AUC(infinity) is calculated as (AUC[infinity] minus AUC[last] divided by AUC[infinity]) multiplied by 100.
Elimination half-life period (t1/2) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36 and 48 hours post-dose of study medication
  Elimination half-life associated with the terminal slope (lambda[z]) of the semi logarithmic drug concentration-time curve, calculated as 0.693/lambda (z).
Terminal slope (Lambda [z]) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36 and 48 hours post-dose of study medication
  Terminal slope is defined by first-order rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Time to Last Quantifiable Serum Concentration (T[last]) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36 and 48 hours post-dose of study medication
  The T(last) is the time to reach last quantifiable serum concentration.
Relative Bioavailability of Tapentadol (F[rel]) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36 and 48 hours post-dose of study medication
  The F(rel) of tapentadol is calculated as the Area Under the Serum Concentration-Time Curve (AUC) and Cmax ratios of the two Treatments(that is, treatment effect).

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical R&D, L.L.C Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical R&D, L.L.C
Locations (1):
- Lincoln, Nebraska, United States

REFERENCES:
- See also: A Pivotal Study to Evaluate the Bio-equivalence of the Tapentadol Extended-Release (ER) Tamper-resistant Formulation (TRF) Tablet to the Current Tapentadol ER Prolonged-release 2 (PR2) Tablet — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=3008&filename=CR100456_CSR.pdf